CLINICAL TRIAL: NCT07169019
Title: Gut Microbiome Changes and Clinical Impact Induced by Treatment of Newly Diagnosed Psoriasis Patients With Probiotics and Methotrexate: a Pilot Study
Brief Title: Microbiome and Clinical Response to Probiotics and Methotrexate in Early Psoriasis: a Pilot Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa Gamaleldin Aboulela, Associate Professor of Microbiology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E/C. S/N. T24/2025
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis (PsO)
Keywords: Psoriasis; gut microbiome; methotrexate; probiotics
MeSH Terms: conditions — Psoriasis | interventions — Probiotics; Methotrexate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics and methotrexate group (Experimental): Patients will receive weekly oral methotrexate 15-25 mg/week, along with an oral daily dose of probiotics.
  Interventions: Drug: Probiotics and methotrexate
- Methotrexate group (Active Comparator): Patients will receive weekly oral methotrexate 15-25 mg/week.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Probiotics and methotrexate — weekly oral methotrexate 15-25 mg/week, along with an oral daily dose of probiotics.
  Arms: Probiotics and methotrexate group
Drug: Methotrexate — weekly oral methotrexate 15-25 mg/week
  Arms: Methotrexate group

SUMMARY:
The goal of this clinical trial is to learn if probiotics work to improve the response of psoriatic patients to methotrexate treatment in adults. It will also learn about the beneficial effect of probiotics on the gut microbiota of psoriatic patients treated with methotrexate. The main questions it aims to answer are:

Do probiotics enhance the reduction of disease burden in psoriatic patients under methotrexate treatment? Do probiotics increase the beneficial gut bacteria and decrease the harmful gut bacteria in psoriatic patients under methotrexate treatment? Researchers will compare probiotics intake along with methotrexate to methotrexate alone to see if probiotics work to enhance the reduction of the severity of psoriasis in patients treated by methotrexate and whether the addition of probiotics will improve their gut health.

Participants will:

Take a daily dose of probiotics with a weekly dose of methotrexate or only a weekly dose of methotrexate for 4 months.

Give daily feedback to the researchers about their probiotic intake and their dietary intake.

Visit the clinic after 1 and 2 weeks of beginning treatment and then once every 4 weeks for checkups and tests.

DETAILED DESCRIPTION:
This study aims to identify the changes in gut microbiome and the clinical impact induced by treatment of newly diagnosed psoriasis patients with probiotics and methotrexate, compared to the standard first line treatment with methotrexate alone.

Methods

1. Collection of demographic and clinical data:

   * Data about the full medical history will be collected for all patients (including name, age, sex, history of the disease, duration of illness, association with other autoimmune diseases like vitiligo, diabetes type 1, etc).
   * Data about the results of full clinical examination of all patients will be collected.
   * Data about the clinical assessment of the severity of Psoriasis will be collected as indicated by the Psoriasis Activity and Severity Index (PASI) score (which is a quantitative rating score for measuring the severity of psoriatic lesions based on area coverage and plaque appearance). PASI score will be calculated before treatment and every month during treatment. (Appendix 1)
   * Data about base line pretreatment laboratory investigations will be collected: CBC, liver and renal function test.
   * Data about follow up lab investigations will be collected:

     * CBC at week 2 and week 4 after treatment and every month thereafter.
     * Liver function tests at week 2 after treatment and every month thereafter.
     * Renal function tests at week 1 after treatment and every month thereafter.
2. Stool samples will be collected from every participant at baseline (before the start of treatment) and at the end of the 16th week of treatment (at the efficacy of treatment assessment visit). Samples will be stored in sterile screw-capped tubes, and kept at -80 ºC, till the time of subsequent experiments.
3. Total DNA will be isolated from stool samples using QIAamp DNA Stool Mini Kit following the manufacturer's instructions.
4. Illumina Next generation sequencing: The microbiota composition will be determined by amplification of the V3 and V4 hypervariable regions of the 16S rRNA gene using universal primers with Illumina compatible adaptors.

   * 16S Metagenomic Sequencing Library will be prepared according to the Illumina Protocol.
   * Bioinformatic analysis of 16S rRNA amplicon sequencing data will be performed for classification of reads at taxonomic levels.
5. Changes in microbiome profiles of participants will be determined and correlated with the clinical outcome of treatment.
6. Statistical analysis: The obtained results from the cases the controls will be statistically analyzed using the appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with chronic plaque psoriasis.

Exclusion Criteria:

* • Psoriatic patients who used systemic treatments at least 3 months before the study, with the exception of acetritin use, in the last 3 years.

  * Patients who have skin infection or other skin or autoimmune diseases such as SLE, Lichen planus, Dermatomyositis and Vitiligo, by history and examination.
  * Pregnant or Lactating mothers.
  * Patients with any contraindication to methotrexate treatment.
  * Patients who develop any adverse reaction during systemic treatment with methotrexate that necessitates cessation of treatment before the 16th week, such as bone marrow suppression as indicated by CBC, elevated liver enzymes, or severe GIT upset.
  * Patients with low intellectual capacity, uneducated patients, or patients unable or unwilling to provide daily feedback about their compliance to the provided probiotics treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To identify the changes in gut microbiome and the clinical impact induced by treatment of newly diagnosed psoriasis patients with probiotics and methotrexate, compared to the standard treatment with methotrexate alone. | One year
  The composition of gut microbiota before the start of treatment and after the end of the treatment course will be determined by analysis of a stool sample from each participant by illumina Next generation sequencing and 16S Metagenomics bioinformatics analysis of data to identify microbial taxa in the samples.
  The clinical impact induced by treatment of newly diagnosed psoriatic patients with probiotics and methotrexate or methotrxate alone will be determined by the calculation of PASI score before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ezzeldin A. Saleh, PhD, Study Chair — Medical Research Institute, Alexandria University; Gamaleldin A. Elsawaf, PhD, Study Director — Medical Research Institute, Alexandria University; Mohamed A. Alqasem, MSc, Principal Investigator — Medical Research Institute, Alexandria University
Locations (1):
- Medical Research Institute, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mu Q, Kirby J, Reilly CM, Luo XM. Leaky Gut As a Danger Signal for Autoimmune Diseases. Front Immunol. 2017 May 23;8:598. doi: 10.3389/fimmu.2017.00598. eCollection 2017. PMID 28588585
- [Result] Strati F, Lattanzi G, Amoroso C, Facciotti F. Microbiota-targeted therapies in inflammation resolution. Semin Immunol. 2022 Jan;59:101599. doi: 10.1016/j.smim.2022.101599. Epub 2022 Mar 15. PMID 35304068
- [Result] Celoria V, Rosset F, Pala V, Dapavo P, Ribero S, Quaglino P, Mastorino L. The Skin Microbiome and Its Role in Psoriasis: A Review. Psoriasis (Auckl). 2023 Oct 26;13:71-78. doi: 10.2147/PTT.S328439. eCollection 2023. PMID 37908308
- [Result] Navarro-Lopez V, Martinez-Andres A, Ramirez-Bosca A, Ruzafa-Costas B, Nunez-Delegido E, Carrion-Gutierrez MA, Prieto-Merino D, Codoner-Cortes F, Ramon-Vidal D, Genoves-Martinez S, Chenoll-Cuadros E, Perez-Orquin JM, Pico-Monllor JA, Chumillas-Lidon S. Efficacy and Safety of Oral Administration of a Mixture of Probiotic Strains in Patients with Psoriasis: A Randomized Controlled Clinical Trial. Acta Derm Venereol. 2019 Nov 1;99(12):1078-1084. doi: 10.2340/00015555-3305. PMID 31453631
- [Result] Amatore F, Villani AP, Tauber M, Viguier M, Guillot B; Psoriasis Research Group of the French Society of Dermatology (Groupe de Recherche sur le Psoriasis de la Societe Francaise de Dermatologie). French guidelines on the use of systemic treatments for moderate-to-severe psoriasis in adults. J Eur Acad Dermatol Venereol. 2019 Mar;33(3):464-483. doi: 10.1111/jdv.15340. Epub 2019 Feb 22. PMID 30793796
- [Result] Brenchley JM, Douek DC. Microbial translocation across the GI tract. Annu Rev Immunol. 2012;30:149-73. doi: 10.1146/annurev-immunol-020711-075001. Epub 2012 Jan 3. PMID 22224779
- [Result] Reali E, Caliceti C, Lorenzini A, Rizzo P. The Use of Microbial Modifying Therapies to Prevent Psoriasis Exacerbation and Associated Cardiovascular Comorbidity. Inflammation. 2024 Feb;47(1):13-29. doi: 10.1007/s10753-023-01915-1. Epub 2023 Nov 13. PMID 37953417
- [Result] Polak K, Bergler-Czop B, Szczepanek M, Wojciechowska K, Fratczak A, Kiss N. Psoriasis and Gut Microbiome-Current State of Art. Int J Mol Sci. 2021 Apr 26;22(9):4529. doi: 10.3390/ijms22094529. PMID 33926088
- [Result] Vicic M, Kastelan M, Brajac I, Sotosek V, Massari LP. Current Concepts of Psoriasis Immunopathogenesis. Int J Mol Sci. 2021 Oct 26;22(21):11574. doi: 10.3390/ijms222111574. PMID 34769005